CLINICAL TRIAL: NCT01485991
Title: Phase III in Partial and Null Responders
Brief Title: TMC435HPC3001 - An Efficacy, Safety and Tolerability Study for TMC435 vs Telaprevir in Combination With PegINFα-2a and Ribavirin in Chronic Hepatitis C Patients Who Were Null or Partial Responders to Prior PegINFα-2a and Ribavirin Therapy
Acronym: ATTAIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR100677; TMC435HPC3001 (Other: Janssen R&D Ireland)
Record Dates: First submitted 2011-11-25; First posted 2011-12-06 (Estimated); Results first posted 2015-04-10 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-03

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; TMC435HPC3001; TMC435; Hepatitis C Virus (HCV); HEP C; Genotype 1; Treatment experienced; Null responders; Partial responders
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TMC435/PR (Experimental)
  Interventions: Drug: TMC435
- TVR/PR (Active Comparator)
  Interventions: Drug: TVR

INTERVENTIONS:
Drug: TMC435 — TMC435 Type=exact number, unit=mg, number=150, form=capsule, route=oral use. TVR placebo Form=tablet, route=oral use. TMC435 capsule is taken once daily in addition to 2 TVR placebo tablets 3 times a day for 12 weeks, and peginterferon alfa-2a and ribavirin for 48 weeks.
  Arms: TMC435/PR
Drug: TVR — TVR Type=exact number, unit=mg, number=375, form=tablet, route=oral use. TMC435 placebo Form=capsule, route=oral use. 2 TVR tablets are taken 3 times a day together with 150 mg TMC435 placebo capsule once daily for 12 weeks, in addition to peginterferon alfa-2a and ribavirin for 48 weeks
  Arms: TVR/PR

SUMMARY:
The purpose of this study is to demonstrate the efficacy of TMC435 in combination with peginterferon (PegIFN) + ribavirin (RBV) by means of establishing its non- inferiority compared to an approved regimen of telaprevir + PegIFN + RBV in patients who have previously failed PegIFN.

DETAILED DESCRIPTION:
This study is a randomized (study drug assigned by chance like flipping a coin), double-blind (neither physician nor patient knows the name of the assigned drug), double-dummy (patients receive both active and inactive pills also called placebo), 2-arm, multicenter Phase III clinical study in adult treatment experienced Chronic Hepatitis C (CHC) genotype-1 infected patients who failed to respond during at least 1 previous course of PegINFα-2a/ RBV therapy. The purpose of the trial is to study the efficacy of TMC435 in combination with PegINFα-2a and RBV for 48 weeks of treatment compared to the approved regimen of telaprevir in combination with PegINFα-2a and RBV for 48 weeks of treatment. The study will consist of a screening period (maximum 6 weeks), treatment period (48 weeks) and post-treatment period (until 72 weeks after the start of treatment). For the first 12 weeks one group of patients will take TMC435 and TVR placebo, plus PegINFα-2a and RBV. The other group will take TMC435 placebo and TVR, plus PegINFα-2a and RBV. After 12 weeks, patients in both arms will only take PegINFα-2a and RBV up to week 48. After patients stop taking study medication, they will continue to go to the doctor's office for study visits until a total of 72 weeks after they start study treatment. Patients will be monitored for safety throughout the study. Study assessments at each study visit may include, but are not limited to: blood and urine collection for testing, electrocardiogram (ECG) assessments (a measurement of the electrical activity of your heart), patient questionnaires, and physical examinations.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have had a liver biopsy before screening (or between the screening and baseline visit), unless patient cannot undergo such a procedure or has evidence of portal hypertension not associated with cirrhosis. For patients who had a liver biopsy performed more than 2 years prior to screening or without a biopsy (because of a contraindication or portal hypertension), a non-invasive staging assessment needs to be available. Non-invasive staging assessments include FibroScan, MR-Elastography, or FibroTest/FibroSure and must not be older than 6 months prior to screening
* Chronicity of hepatitis C virus (HCV) infection, as confirmed by one or both of the following: presence of anti-HCV antibody and/or HCV ribonucleic acid (RNA) at least 6 months prior to the screening visit and/or presence of fibrosis on biopsy
* Genotype 1 HCV infection with plasma HCV RNA of >10,000 IU/mL (both confirmed at screening)
* Patient must have had at least 1 documented previous course of treatment with PegINFα-2a or PegINFα-2b in combination with ribavirin (RBV) (at least 12 weeks for null responder and 20 weeks for partial responder)

Exclusion Criteria:

* Hepatic decompensation (impaired functioning of the liver), as indicated by significant laboratory abnormalities or other active diseases
* Infection with Human Immunodeficiency Virus (HIV) or non genotype 1 hepatitis C
* Liver disease not related to hepatitis C infection
* Previous chronic hepatitis C treatment, other than PegIFN and RBV

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 771 (Actual)
Dates: Start 2012-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Limited Clinical Trial, Study Director — Tibotec Pharmaceutical Limited
Locations (137):
- United States (32):
  - Bakersfield, California
  - San Diego, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Jacksonville, Florida
  - Orlando, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Crestview Hills, Kentucky
  - New Orleans, Louisiana
  - Chevy Chase, Maryland
  - Jackson, Mississippi
  - Tupelo, Mississippi
  - Kansas City, Missouri
  - Missoula, Montana
  - Newark, New Jersey
  - New York, New York
  - Rochester, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Allentown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Arlington, Texas
  - Houston, Texas
  - Odessa, Texas
  - San Antonio, Texas
  - Falls Church, Virginia
  - Bellevue, Washington
  - Seattle, Washington
- Argentina (2):
  - Buenos Aires
  - Rosario, Santa Fe
- Australia (8):
  - Darlinghurst
  - Greenslopes
  - Kingswood
  - Melbourne
  - Parkville - Vic
  - Perth
  - Sydney
  - Woolloongabba
- Austria (2):
  - Linz
  - Vienna
- Belgium (4):
  - Brussels
  - Haine-Saint-Paul, La Louviere
  - Leuven
  - Liège
- Brazil (4):
  - Campinas
  - Ribeirão Preto
  - Salvador
  - São Paulo
- Bulgaria (2):
  - Sofia
  - Varna
- Canada (5):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Toronto, Ontario
  - Montreal, Quebec
- Czechia (4):
  - Brno
  - Karlovy Vary
  - Pilsen
  - Prague
- Denmark (3):
  - Copenhagen
  - Hvidovre
  - Odense
- France (7):
  - Grenoble
  - Lyon
  - Marseille
  - Nice
  - Paris
  - Pessac
  - Vandœuvre-lès-Nancy
- Germany (12):
  - Berlin
  - Frankfurt
  - Freiburg im Breisgau
  - Hamburg
  - Hanover
  - Heidelberg
  - Kiel
  - Mainz
  - München
  - Stuttgart
  - Ulm
  - Würzburg
- Greece (3):
  - Alexandroupoli
  - Athens
  - Larissa
- Hungary (5):
  - Budapest
  - Debrecen
  - Kaposvár
  - Pécs
  - Szeged
- Israel (6):
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
  - Safed
  - Tel Aviv
- Norway (4):
  - Fredrikstad
  - Nordbyhagen
  - Stavanger
  - Tromsø
- Poland (8):
  - Bydgoszcz
  - Chorzów
  - Kielce
  - Lodz
  - Lublin
  - Mysłowice
  - Racibórz
  - Warsaw
- Portugal (2):
  - Lisbon
  - Porto
- Santurce, Puerto Rico
- Romania (4):
  - Bucharest
  - Constanța
  - Iași
  - Timișoara
- Spain (5):
  - Barcelona
  - Madrid
  - Santander
  - Seville
  - Valencia
- Sweden (5):
  - Gothenburg
  - Lund
  - Malmo
  - Örebro
  - Stockholm
- Switzerland (3):
  - Lugano
  - Sankt Gallen
  - Zurich
- United Kingdom (6):
  - Glasgow
  - Leeds
  - London
  - Newcastle upon Tyne
  - Plymouth
  - Southampton

REFERENCES:
- [Derived] Reddy KR, Zeuzem S, Zoulim F, Weiland O, Horban A, Stanciu C, Villamil FG, Andreone P, George J, Dammers E, Fu M, Kurland D, Lenz O, Ouwerkerk-Mahadevan S, Verbinnen T, Scott J, Jessner W. Simeprevir versus telaprevir with peginterferon and ribavirin in previous null or partial responders with chronic hepatitis C virus genotype 1 infection (ATTAIN): a randomised, double-blind, non-inferiority phase 3 trial. Lancet Infect Dis. 2015 Jan;15(1):27-35. doi: 10.1016/S1473-3099(14)71002-3. Epub 2014 Dec 5. PMID 25482330

RESULTS

PARTICIPANT FLOW:
Groups:
- Simeprevir+Placebo+Peginterferon Alfa-2a+Ribavirin: Simeprevir (TMC435) 150 milligram (mg) capsule, orally, once daily for 12 weeks, along with 2 telaprevir (TVR) matched placebo tablets 3 times a day for 12 weeks, and peginterferon alfa-2a and ribavirin for 48 weeks.
- Telaprevir+Placebo+Peginterferon Alfa-2a+Ribavirin: 2 Telaprevir (TVR) tablets, orally, 3 times a day along with 150 mg TMC435 matched placebo capsule once daily for 12 weeks, in addition to peginterferon alfa-2a and ribavirin for 48 weeks.
Period: Overall Study
Arm/Group | Simeprevir+Placebo+Peginterferon Alfa-2a+Ribavirin | Telaprevir+Placebo+Peginterferon Alfa-2a+Ribavirin
Started | 385 | 386
Treated | 379 | 384
Completed | 353 | 350
Not Completed | 32 | 36
Not completed — Adverse Event | 0 | 4
Not completed — Lost to Follow-up | 13 | 10
Not completed — Withdrawal by Subject | 13 | 20
Not completed — randomized but not treated | 6 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants who took at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Simeprevir+Placebo+Peginterferon Alfa-2a+Ribavirin | Telaprevir+Placebo+Peginterferon Alfa-2a+Ribavirin | Total
Number analyzed (Participants) | 379 | 384 | 763
Age, Continuous [Median (Full Range); unit: years] | 50 [18 to 69] | 52 [20 to 69] | 51 [18 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 161 | 297
  Male | 243 | 223 | 466

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After the Planned End of Treatment (SVR12)
Description: Participants are considered to have reached SVR12 if both conditions below are met: 1) HCV RNA levels less than (<) 25 International unit per milliliter (IU/mL) undetectable; 2) HCV RNA levels <25 IU/mL undetectable or HCV RNA levels <25 IU/mL detectable.
Time Frame: 12 Weeks After the Planned End of Treatment (EOT: Week 48)
Population: Intent-to-treat (ITT) population included all randomized participants who took at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Simeprevir+Placebo+Peginterferon Alfa-2a+Ribavirin | Telaprevir+Placebo+Peginterferon Alfa-2a+Ribavirin
Number analyzed (Participants) | 379 | 384
percentage of participants | 53.6 | 54.7
Statistical Analysis 1: Comparison: Simeprevir+Placebo+Peginterferon Alfa-2a+Ribavirin vs Telaprevir+Placebo+Peginterferon Alfa-2a+Ribavirin; Test type: Superiority or Other; p = 0.001, Stratified Cochran-Mantel-Haenszel — based on the asymptotic distribution of the generalized Cochran-Mantel-Haenszel statistic controlling for stratification factors, using a non-inferiority margin of 12 percent; Difference in proportions = -1.1, 95% CI 2-sided [-7.8 to 5.5]

2. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks After the Planned End of Treatment (SVR24)
Description: Participants are considered to have reached SVR24 if both conditions below are met: 1) HCV RNA levels less than <25 International unit per milliliter (IU/mL) undetectable (at the actual end of treatment);2) HCV RNA levels <25 IU/mL undetectable or HCV RNA levels <25 IU/mL detectable (24 weeks after the planned EOT).
Time Frame: 24 Weeks After the Planned EOT (Week 48)
Population: ITT population included all randomized participants who took at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Simeprevir+Placebo+Peginterferon Alfa-2a+Ribavirin | Telaprevir+Placebo+Peginterferon Alfa-2a+Ribavirin
Number analyzed (Participants) | 379 | 384
percentage of participants | 53.3 | 55.2

3. Secondary Outcome: Percentage of Participants With Viral Relapse
Description: Participants are considered to have a viral relapse if both conditions as specified are met: 1) <25 IU/mL undetectable HCV RNA at the actual end of study drug treatment; 2) confirmed HCV RNA greater than or equal to (>=) 25 IU/mL during follow-up.
Time Frame: End of Treatment (Week 48) up to Follow-up Period (until Week 72)
Population: ITT population included all randomized participants who took at least 1 dose of study drug. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Simeprevir+Placebo+Peginterferon Alfa-2a+Ribavirin | Telaprevir+Placebo+Peginterferon Alfa-2a+Ribavirin
Number analyzed (Participants) | 246 | 256
percentage of participants | 17.9 | 16.4

ADVERSE EVENTS:
Time Frame: Baseline up to Follow-up (Week 72)
Arm/Group | Simeprevir+Placebo+Peginterferon Alfa-2a+Ribavirin | Telaprevir+Placebo+Peginterferon Alfa-2a+Ribavirin
Serious Adverse Events (participants affected / at risk) | 22/379 | 54/384
Other Adverse Events (participants affected / at risk) | 349/379 | 369/384
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Simeprevir+Placebo+Peginterferon Alfa-2a+Ribavirin (N=379) | Telaprevir+Placebo+Peginterferon Alfa-2a+Ribavirin (N=384)
Anaemia (Blood and lymphatic system disorders) | 2 | 16
Neutropenia (Blood and lymphatic system disorders) | 2 | 3
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 4
Appendicitis (Infections and infestations) | 2 | 1
Acute sinusitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Superinfection (Infections and infestations) | 1 | 0
Candidiasis (Infections and infestations) | 0 | 1
Impetigo (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia legionella (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Critical illness polyneuropathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Mononeuropathy (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0
Drug rash with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2
Thrombophlebitis (Vascular disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 0
Fatigue (General disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Chemical peritonitis (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Simeprevir+Placebo+Peginterferon Alfa-2a+Ribavirin (N=379) | Telaprevir+Placebo+Peginterferon Alfa-2a+Ribavirin (N=384)
Fatigue (General disorders) | 132 | 155
Pyrexia (General disorders) | 86 | 101
Asthenia (General disorders) | 80 | 69
Influenza like illness (General disorders) | 64 | 66
Chills (General disorders) | 22 | 40
Injection site erythema (General disorders) | 14 | 27
Pruritus (Skin and subcutaneous tissue disorders) | 142 | 179
Rash (Skin and subcutaneous tissue disorders) | 66 | 100
Dry skin (Skin and subcutaneous tissue disorders) | 39 | 30
Alopecia (Skin and subcutaneous tissue disorders) | 33 | 59
Anaemia (Blood and lymphatic system disorders) | 95 | 157
Neutropenia (Blood and lymphatic system disorders) | 82 | 78
Thrombocytopenia (Blood and lymphatic system disorders) | 40 | 46
Nausea (Gastrointestinal disorders) | 74 | 110
Diarrhoea (Gastrointestinal disorders) | 51 | 60
Dyspepsia (Gastrointestinal disorders) | 25 | 29
Abdominal pain upper (Gastrointestinal disorders) | 24 | 25
Vomiting (Gastrointestinal disorders) | 23 | 36
Constipation (Gastrointestinal disorders) | 21 | 10
Abdominal pain (Gastrointestinal disorders) | 11 | 22
Dry mouth (Gastrointestinal disorders) | 11 | 25
Anorectal discomfort (Gastrointestinal disorders) | 10 | 32
Anal pruritus (Gastrointestinal disorders) | 9 | 42
Haemorrhoids (Gastrointestinal disorders) | 6 | 38
Headache (Nervous system disorders) | 103 | 120
Dizziness (Nervous system disorders) | 26 | 43
Dysgeusia (Nervous system disorders) | 15 | 36
Insomnia (Psychiatric disorders) | 53 | 73
Depression (Psychiatric disorders) | 35 | 20
Mood altered (Psychiatric disorders) | 35 | 32
Cough (Respiratory, thoracic and mediastinal disorders) | 66 | 53
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30 | 40
Myalgia (Musculoskeletal and connective tissue disorders) | 47 | 63
Arthralgia (Musculoskeletal and connective tissue disorders) | 41 | 45
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 30
Decreased appetite (Metabolism and nutrition disorders) | 54 | 64
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 28
Urinary tract infection (Infections and infestations) | 12 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.